CLINICAL TRIAL: NCT00590044
Title: Basal Insulin in the Management of Patients With Diabetic Ketoacidosis
Brief Title: Basal Insulin in the Management of Patients With Diabetic Ketoacidosis (DKA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00005062a
Record Dates: First submitted 2007-12-28; First posted 2008-01-10 (Estimated); Results first posted 2009-04-30 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Diabetic Ketoacidosis
Keywords: Diabetic ketoacidosis; insulin therapy; DKA
MeSH Terms: conditions — Diabetic Ketoacidosis | interventions — Insulin Glargine; insulin glulisine; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin glargine+glulisine (Experimental): Daily insulin glargine + glulisine before meals
  Interventions: Drug: insulin glargine+ glulisine
- Split-mixed NPH + Regular insulin (Active Comparator): Split-mixed NPH + Regular insulin twice daily
  Interventions: Drug: NPH + Regular insulin

INTERVENTIONS:
Drug: insulin glargine+ glulisine — Daily insulin glargine + glulisine before meals
  Other Names: glargine (Lantus) + glulisine (Apidra)
  Arms: Insulin glargine+glulisine
Drug: NPH + Regular insulin — Split-mixed NPH + Regular insulin twice daily
  Other Names: Isophane Insulin(NPH); Intermediate acting Insulin (NPH)
  Arms: Split-mixed NPH + Regular insulin

SUMMARY:
The study is a multicenter, randomized controlled trial to compare the safety and efficacy of insulin analogs and human insulins both during acute intravenous treatment and during the transition to subcutaneous insulin in patients with diabetic ketoacidosis (DKA).

DETAILED DESCRIPTION:
Diabetic ketoacidosis (DKA) is the most serious emergency in patients with diabetes. With an estimated 100,000 admissions per year in the United States, DKA is also the leading cause of death in children with type 1 diabetes, and accounts for a significant proportion of admissions in adult patients with type 1 and type 2 diabetes. The mainstay in the treatment of DKA involves the continuous intravenous (IV) infusion of regular insulin or the frequent subcutaneous (SC) injections of regular or rapid-acting insulin analogs. Multiple studies have reported successful protocols for insulin administration during the acute management of DKA, but they have failed to address the transition phase from IV to SC maintenance insulin regimen. The American Diabetes Association (ADA) position statement recommends the use of split-mixed insulin combination of regular and intermediate-acting insulin (NPH). This regimen, however, are associated with a high rate of hyperglycemia shortly after discontinuation of IV insulin and a risk of hypoglycemia during the hospital stay. Recently, the long-acting "basal" insulin glargine (Lantus®, Sanofi Aventis Pharmaceuticals) has been shown to facilitate glycemic control with lower rate of hypoglycemic events than intermediate-acting insulin in subjects with type 1 and type 2 diabetes. This study aims i) to determine the effects of giving a dose of glargine insulin shortly after starting an intravenous insulin infusion on glycemic control, time to resolve DKA, and rate of hypoglycemia in patients with DKA, and ii) to compare the safety and efficacy of basal/bolus (glargine/glulisine) insulin versus the standard split-mixed insulin regimen of NPH and regular insulin after the resolution of DKA. The hypothesis is that basal (lantus®) insulin as compared to NPH insulin shortly after the start of insulin infusion will improve inpatient glycemic control in patients with DKA.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Grady Memorial Hospital who meet diagnosis criteria of DKA and who are willing to participate in the study protocol will be considered candidates for inclusion into the study.
* Diagnostic Criteria for DKA: Blood glucose > 250 mg/dL, arterial or venous phenol hydroxylase (pH) < 7.3, serum bicarbonate < 18 milliequivalent/L, and moderate to severe ketonemia (acetoacetate ≥ 1:4 or βeta-hydroxybutyrate > 3 mmol).

Exclusion Criteria:

* Hemodynamic instability (MAP < 50 or patients requiring pressor)
* Significant identifiable medical or surgical illness, including but not limited to: acute myocardial infarction, congestive heart failure; respiratory failure requiring mechanical ventilation; acute or chronic renal insufficiency (serum creatinine > 3.0 mg/dl); end stage liver failure, and cirrhosis.
* Patients with dementia or persistent altered mental status that would prevent collection of consent form and reliable information.
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University SOM; Sidney Jones, MD, Study Chair — University of Minnesota
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - University of Minnesota School of Medicine, Minneapolis, Minnesota

REFERENCES:
- [Result] Umpierrez GE, Jones S, Smiley D, Mulligan P, Keyler T, Temponi A, Semakula C, Umpierrez D, Peng L, Ceron M, Robalino G. Insulin analogs versus human insulin in the treatment of patients with diabetic ketoacidosis: a randomized controlled trial. Diabetes Care. 2009 Jul;32(7):1164-9. doi: 10.2337/dc09-0169. Epub 2009 Apr 14. PMID 19366972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at Grady Memorial Hospital, Atlanta, Georgia, and at Hennepin County Medical Center, Minneapolis, Minnesota
Pre-assignment Details: A total of 74 patients with DKA were randomly assigned. Of them, 6 were excluded because 4 withdrew consent before or shortly after initiation of insulin therapy, one patient received glargine insulin before resolution of DKA, and one patient was treated with IV aspart insulin instead of regular insulin. The remaining 68 were included in analysis
Groups:
- Glargine (Lantus) + Glulisine: Daily insulin glargine (Lantus) + glulisine (Apidra) before meals
- NPH + Regular: Split-mixed NPH + Regular insulin twice daily
Period: Overall Study
Arm/Group | Glargine (Lantus) + Glulisine | NPH + Regular
Started | 38 | 36
Completed | 34 | 34
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — wrong insulin arm assigned | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glargine (Lantus) + Glulisine | NPH + Regular | Total
Number analyzed (Participants) | 38 | 36 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 36 | 74
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (12) | 38 (12) | 38.5 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 24 | 24 | 48
Region of Enrollment [Number; unit: participants]
  United States | 38 | 36 | 74

OUTCOME MEASURES:

1. Primary Outcome: Number of Hypoglycemia Episodes After the Transition Period From Intravenous Insulin to Subcutaneous Insulin Between 2 Treatment Groups
Description: To determine the safety of the two treatments the number of hypoglycemia episodes that occurred between the 2 groups are measured from the time of transitioning to subcutaneous insulin to day 5. The hypoglycemia events are defined as blood glucose levels <70 mg/dL. The results were obtained from the citation Umpierrez GE, Jones S, Smiley D, Mulligan P, Keyler T, Temponi A, Semakula C, Umpierrez D, Peng L, Cerón M, Robalino G. Insulin analogs versus human insulin in the treatment of patients with diabetic ketoacidosis: a randomized controlled trial. Diabetes Care. 2009 Jul;32(7):1164-9. doi: 10.2337/dc09-0169. Epub 2009 Apr 14. PubMed ID: 19366972.
Time Frame: 5 days after transitioning to subcutaneous insulin
Measure: Number; unit: number of hypoglycemia episodes
Arm/Group | Insulin Glargine+Glulisine | Split-mixed NPH + Regular Insulin
Number analyzed (Participants) | 34 | 34
number of hypoglycemia episodes | 8 | 26

2. Secondary Outcome: Mean Daily Blood Glucose Concentration Between the Two Groups After the Resolution of Ketoacidosis and Transition to Subcutaneous Insulin
Description: The primary outcome during the subcutaneous (SC) period (the primary outcome measurement) was to determine differences in glycemic control as measured by mean daily blood glucose(BG) concentration between treatment groups. The results were obtained from the citation Umpierrez GE, Jones S, Smiley D, Mulligan P, Keyler T, Temponi A, Semakula C, Umpierrez D, Peng L, Cerón M, Robalino G. Insulin analogs versus human insulin in the treatment of patients with diabetic ketoacidosis: a randomized controlled trial. Diabetes Care. 2009 Jul;32(7):1164-9. doi: 10.2337/dc09-0169. Epub 2009 Apr 14. PubMed Identification (ID): 19366972.
Time Frame: Day1 - Day5 after the resolution of ketoacidosis and transition to subcutaneous insulin
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- NPH + Regular: Split-mixed Isophane (NPH) + Regular insulin twice daily
Arm/Group | Glargine (Lantus) + Glulisine | NPH + Regular
Number analyzed (Participants) | 34 | 34
mg/dl
  Day 1 | 213 (76) | 188 (61)
  Day 2 | 220 (61) | 206 (71)
  Day 3 | 180 (80) | 207 (86)
  Day 4 | 158 (44) | 211 (63)
  Day 5 | 124 (41) | 190 (45)

3. Secondary Outcome: Mean Blood Glucose Concentration in mg/dL While on the Insulin Drip Among the 2 Groups
Description: To determine the differences in glycemic control as measured by differences in the mean daily blood glucose levels between treatment groups (insulin drip with regular insulin vs glulisine insulin) during the acute phase of diabetic ketoacidosis(DKA) before transitioning to subcutaneous insulin. The results were obtained from the citation Umpierrez GE, Jones S, Smiley D, Mulligan P, Keyler T, Temponi A, Semakula C, Umpierrez D, Peng L, Cerón M, Robalino G. Insulin analogs versus human insulin in the treatment of patients with diabetic ketoacidosis: a randomized controlled trial. Diabetes Care. 2009 Jul;32(7):1164-9. doi: 10.2337/dc09-0169. Epub 2009 Apr 14. PubMed ID: 19366972.
Time Frame: up to 20 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Glargine (Lantus) + Glulisine | NPH + Regular
Number analyzed (Participants) | 34 | 34
mg/dL | 153 (61) | 185 (58)

4. Secondary Outcome: Difference in Time in Hours to Resolution of DKA Between the 2 Groups
Description: The mean duration of treatment until resolution of ketoacidosis is measured and compared between the 2 groups. The DKA was considered resolved when blood glucose was 250 mg/dl, the serum bicarbonate level was <18 mmol/l, and venous phenol hydroxylase (pH) was 7.30. The results were obtained from the citation Umpierrez GE, Jones S, Smiley D, Mulligan P, Keyler T, Temponi A, Semakula C, Umpierrez D, Peng L, Cerón M, Robalino G. Insulin analogs versus human insulin in the treatment of patients with diabetic ketoacidosis: a randomized controlled trial. Diabetes Care. 2009 Jul;32(7):1164-9. doi: 10.2337/dc09-0169. Epub 2009 Apr 14. PubMed ID: 19366972.
Time Frame: up to 20 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Glargine (Lantus) + Glulisine | NPH + Regular
Number analyzed (Participants) | 34 | 34
hours | 8.9 (4.7) | 10.5 (6.3)

ADVERSE EVENTS:
Time Frame: The adverse event data are collected from the time of admission to day 5 after the resolution of diabetic ketoacidosis (DKA).
Description: For this study the adverse events of interest were hypoglycemia events where glucose levels are <70 mg/dL and severe hypoglycemia events with glucose level <40 mg/dL. The events were collected from rom the time of admission to day 5 after the resolution of diabetic ketoacidosis (DKA). The rest of the treatments for the patients was standard of care treatment.
Arm/Group | Glargine (Lantus) + Glulisine | NPH + Regular
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/38 | 2/36
Other Adverse Events (participants affected / at risk) | 5/38 | 14/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glargine (Lantus) + Glulisine (N=38) | NPH + Regular (N=36)
Severe Hypoglycemia (Endocrine disorders) | 1 (1) | 2 (2) — Severe hypoglycemia is defined as blood glucose level < 40 mg/dL that required immediate invasive intervention
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glargine (Lantus) + Glulisine (N=38) | NPH + Regular (N=36)
Hypoglycemia (Endocrine disorders) | 5 (8) | 14 (26) — Hypoglycemia is defined as blood glucose level <70 mg/dL

LIMITATIONS AND CAVEATS:
The study included relatively small number of patients. The study also excluded patients with hypovolemic shock, comatose patients and patients who had acute myocardial ischemia, congestive heart failure, end-stage renal or hepatic failure..

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No